CLINICAL TRIAL: NCT06601634
Title: Predictors of Axial Pain Improvement After Anterior Cervical Discectomy and Fusion - Prospective, Observational Study
Brief Title: Predictors of Axial Pain Improvement After Anterior Cervical Discectomy and Fusion
Status: Recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Jan Chrzanowski, MD, Medical University of Warsaw
Other Study IDs: WUMStudy
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Neck Pain; Cervical Spondylosis; Cervical Disc Disease
MeSH Terms: conditions — Neck Pain; Spondylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neck pain is a common, multifactorial condition. In the case of degenerative cervical spinal disease, it can result from changes in the intervertebral discs, muscles, intervertebral joints, or sagittal imbalance. Anterior cervical discectomy and fusion (ACDF) is a currently widely accepted procedure for treating cervical degenerative spine disease, with a high patient satisfaction rate. In the current state of knowledge, it is not used for treating axial neck pain, but rather in cases of discopathy causing spinal myelopathy or cervical radiculopathy, in which neck pain often coexists or predominates. The current literature provides ample evidence of the significant effect of ACDF in improving axial neck pain in the conditions mentioned previously. However, little information exists on which patients achieve improvement. The aim of this prospective study is to analyze the outcomes of ACDF in patients with neck pain and to identify predictors of reduction in axial neck pain after ACDF.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Patients who are qualified for one- or two-level ACDF for the treatment of degenerative cervical pathology

Exclusion Criteria:

* Previous cervical spine surgery
* Previous cervical spine trauma
* Other diseases causing neck pain include rheumatoid arthritis, lupus, polymyalgia rheumatica, myositis, seronegative inflammatory diseases, and fibromyalgia
* Drug abuse
* Myelopathy
* Spinal infection
* VAS neck pain score less than 3 (Inability to achieve an MCID which is calculated as 2.5 for the VAS scale)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to prospectively enroll at least 60 patients who are qualified for one- or two-level ACDF for the treatment of degenerative cervical pathology with significant neck pain, and to identify predictors of the reduction in axial neck pain following surgery.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-17 (Actual); Primary Completion 2027-11-17 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Predictors of the reduction of axial neck pain following ACDF. | On the day of discharge from the hospital, at 6 months, 1 year, 2 years
  Change in VAS neck pain ( visual analog scale), with calculated MCID ( Minimal Clinically Important Difference) as 2.5
Predictors of functional outcomes following ACDF. | On the day of discharge from the hospital, at 6 months, 1 year, 2 years
  Change in NDI ( neck disability index), with calculated MCID as 7.5

SECONDARY OUTCOMES:
Predictors of the reduction of axial neck pain following ACDF in population with predominant neck pain. | On the day of discharge from the hospital, at 6 months, 1 year, 2 years
  Change in VAS neck pain ( visual analog scale), with calculated MCID ( Minimal Clinically Important Difference) as 2.5 in population with predominant neck pain. (VAS neck - VAS arm ≥ 1.0 point)
Predictors of functional outcomes following ACDF in population with predominant neck pain. | On the day of discharge from the hospital, at 6 months, 1 year, 2 years
  Change in NDI ( neck disability index), with calculated MCID as 7.5 in population with predominant neck pain. (VAS neck - VAS arm ≥ 1.0 point)

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Department of Orthopaedics, J. Dietl Specialist Hospital, Krakow, Lesser Poland Voivodeship
  - Department of Neurosurgery, Medical University of Warsaw, Warsaw, Masovian Voivodeship

IPD SHARING:
Plan to Share IPD: Undecided